CLINICAL TRIAL: NCT06136000
Title: Sacral Circumcision Surgery: Comparison of the Effects of Erector Spina Plane Block and Ring Block on Postoperative Pain
Brief Title: S-ESP and Ring Block in Circümcision Surgery (S-ESP: Sacral Erectör Spinae Plane Block).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, Department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY SACRAL ERECTÖR
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pain; Pain, Postoperative
Keywords: erectör spinae plane block; ring block; postoperative analgesia
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SACRAL EREKTÖR SPİNAE PLANE BLOK (Active Comparator)
  Interventions: Other: Sacral erectör spinae plane block
- RİNG BLOCK (Active Comparator)
  Interventions: Other: Ring Block

INTERVENTIONS:
Other: Sacral erectör spinae plane block — Group S will be placed on their side. Asepsis is fifth in the transverse plane under antisepsis standards. high-frequency linear USG probe into the spinous process . The USG probe will be shifted caudally to visualize the first and second median sacral crest. The USG probe is then placed on the second medial It will be placed 3-4 cm lateral to the sacral apex and the mid-sacral apex will be imaged. On the USG screen, from top to bottom, erector spinae muscle, multifidus muscle and sacral intermediate The crest will be displayed. 0.25% bupivacaine will be administered in a total volume of 0.5ml/kg (maximum 20 cc ) by applying negative aspiration with the in-plane technique with a 50 mm Stimuplex A needle.
  Arms: SACRAL EREKTÖR SPİNAE PLANE BLOK
Other: Ring Block — The patient is under general anesthesia. Before the surgical procedure begins, the pediatric surgeon administers 0.5ml/kg (maximum 20cc) 0.25% bupivacaine to the base of the root of the penis with a 25-gauge needle at 3, 6, 9, and 12 o'clock.
  Arms: RİNG BLOCK

SUMMARY:
Although it is not known exactly when and where circumcision was first performed, it is claimed that it was first performed by the Egyptians, according to various beliefs and traditions. Circumcision is the surgical removal of the skin surrounding the glans penis in pediatric male patients and is the most commonly performed surgery in boys (4). Because the foreskin is sensitive and the pain threshold is low, patients experience severe pain in the postoperative period. Various analgesic methods have been developed to reduce this pain. Sacral surgery has started to be used in adult patients in recent years, but there is not enough information about its application in pediatric patients. Sacral erector spinae plane block is on the agenda. While sacral erectör spinae plane block was first applied in gender reassignment and pilonidal sinus surgery in adults, it was also applied to a small extent in hypospadias and anoplasty surgery in pediatric patients. In some studies, circumcision surgery involves the root and distal parts of the penis. It has been emphasized that ring blocks applied with anesthesia also have an analgesic effect. Our aim in this study was to compare the effect of S-ESPB and ring block on postoperative Face, Legs, Movement, Crying, Avocative Behavioral Scale pain scores in pediatric patients undergoing circumcision surgery and to compare the number of patients who required rescue analgesia, the time until the first rescue analgesia, possible complications, and parental satisfaction (a Likert scale will be used).

In this study, we found that sacral erectör spinae plane block is different from the ring block applied in routine practice in circumcision surgery. We think that postoperative analgesic effectiveness will be higher.

Our aim in this study was to compare the effect of sacral erectör spinae plane block and ring block on postoperative Face, Legs, Movement, Crying, Avocative Behavioral Scale pain score in pediatric patients undergoing circumcision surgery and to compare the number of patients who required rescue analgesia secondarily, the time until the first rescue analgesia, possible complications and parental satisfaction (Likert scale will be used).

DETAILED DESCRIPTION:
Our primary hypothesis erectör spinae plane block will be effective in pediatric patients undergoing circumcision surgery. The effect on postoperative pain will be greater than the applied ring block and the Face, Legs, Movement, Crying, Avocative Behavioral Scale pain score will be lower.

Our secondary hypothesis is that the number of patients requiring rescue analgesia and the complications that may occur will be lower in sacral erectör spinae plane block to be applied in circumcision surgery compared to the ring block, and parental satisfaction and the time until the first rescue analgesia will be higher.

Material oath methods: Our study will be carried out within 6 months with 50 patients in the operating room of Konya City Hospital of the University of Health Sciences and the operating room of Harran University Faculty of Medicine Randomization This study was a multicenter prospective study. It was planned and will be carried out as a randomized study. Randomization will be carried out by the sealed envelope method. Patients will be divided into two groups: Group R (patients who underwent Ring block) and Group S (patients who underwent sacral erectör spinae plane block). Since it is a multicenter study, the anesthesia technique will be applied by two different physicians with at least five years of clinical experience and the postoperative results will be recorded by 2 different physicians. These physicians will evaluate patients completely independently and blindly. Written and verbal consent will be obtained from the patient's parents.

Anesthesia Technique and Analgesia Protocol:

Routine anesthesia monitoring and method will be applied to all patients. 22 gauge to patients Intravenous ( IV ) cannulation is provided and 15cc/kg/ h Isotonic fluid will be started. General anesthesia induction 1mg midazolam IV, 2 mg/kg propofol IV, and 1 mcg /kg remifentanil It will be done by giving IV. The patients will be fitted with a laryngeal mask airway (LMA), which we use in routine practice, and will require minimum anesthesia maintenance. alveolar Sevoflurane will be given with a concentration (MAC) value of 1. Before the surgical procedure begins, sacral erectör spinae plane block will be applied to the patients by the anesthesiologist or ring block by the pediatric surgeon. Then circumcision surgery will begin. The same surgical method will be applied to all patients.

At the end of the surgery, we routinely administer 15 mg/kg IV to all patients. Paracetamol will be given. Extubated patients will be transferred to the postanesthetic care unit (PACU) for observation. 0-1-2-4-6 from the time patients are admitted to the PACU until they are discharged from the hospital. Pain levels will be evaluated with the Face, Legs, Movement, Crying, Avocative Behavioral Scale pain scale. Patients with a Face, Legs, Movement, Crying, Avocative Behavioral Scale score of 4 and above will be given 10 mg/kg oral ibuprofen rescue analgesia. The number of patients requiring rescue analgesia, the time until the first rescue analgesia, complications that will develop, and parental satisfaction will be recorded.

sacral erectör spinae plane block with ultrasound guidance Group S will be placed on their side. Asepsis is fifth in the transverse plane under antisepsis standards. high-frequency [(10-15 millihertz ( mHz )] linear ultrasonography probe into the spinous process The ultrasonography probe will be shifted caudally to visualize the first and second median sacral crest. The USG probe is then placed on the second medial It will be placed 3-4 cm lateral to the sacral apex and the mid-sacral apex will be imaged. On the ultrasonography screen, from top to bottom, erector spinae muscle, multifidus muscle and sacral intermediate The crest will be displayed. 0.25% bupivacaine will be administered in a total volume of 0.5ml/kg (maximum 20 cc ) by applying negative aspiration with the in-plane technique with a 50 mm Stimuplex A needle. The process will be applied bilaterally.

Ring Block It is a block that is routinely performed in our clinic by a pediatric surgeon. The patient is under general anesthesia. Before the surgical procedure begins, the pediatric surgeon administers 0.5ml/kg (maximum 20cc) 0.25% bupivacaine to the base of the root of the penis with a 25-gauge needle at 3, 6, 9, and 12 o'clock. local It will be administered under anesthesia.

Primary evaluation criteria are the Face, Legs, Movement, Crying, Avocative Behavioral Scale of pain at rest and movement at 0, 1, 2, 4, and 6 hours after surgery (0-10, 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7- It will be evaluated with 10 = the most severe pain).

Secondary evaluation criteria are the number of patients needing rescue analgesia, the time until the first rescue analgesia, the complications that will develop, and parental satisfaction. The age, weight, height, and surgery duration of the patients in both groups were recorded. Likert evaluation test will be applied for parental satisfaction.

Sample Size:

for circumcision under general anesthesia. patients who will undergo surgery. In the sample size analysis, it was determined that there should be 19 patients for each group with a 95% power rate and an alpha margin of error of 0.05 for comparison of the two groups. The effect used for this calculation is 1.106, based on similar studies, actual power was calculated as 0.955. As a result of the analysis, drop Considering the out rate, it was planned to recruit 25 patients for each group (50 patients in total).

Statistical Analyzes To determine whether the data is normally distributed, the Shapiro Wilks test will be used. Descriptive statistical analyses will be used to evaluate demographic data and data obtained from tests and scales. A paired sample T-test will be used to compare data. Correlation analysis will be used to evaluate the relationship between data. Data will be expressed as mean ± standard deviation and percentage. P <0.05 will be considered statistically significant. In correlation analysis, confidence intervals and p-values will be evaluated according to whether they show a statistically significant or non-significant inverse interaction.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 4-16
* patients with ASA I-II.
* Patients who will receive general anesthesia

Exclusion Criteria:

* Parents and patients who do not want to give consent
* Patients with ASAIII and above
* Patients with a disordered bleeding profile
* Patients using anticoagulants
* Patients with infection in the area to be treated

Ages: 4 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — BOYS WHO WILL BE CIRCUMCISED
Enrollment: 50 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Movement, Crying, Avocative Behavioral Scale | FİVE MONTHS
  Primary evaluation criteria are the Face, Legs, Movement, Crying, Avocative Behavioral Scaleof pain at rest and movement at 0, 1, 2, 4, and 6 hours after surgery (0-10, 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7- It will be evaluated with 10 = the most severe pain).

SECONDARY OUTCOMES:
Postoperative rescue analgesia | FİVE MONTHS
  Secondary evaluation criteria are The number of patients needing rescue analgesia, the time until the first rescue analgesia, the complications that will develop, and parental satisfaction. The age, weight (kilogram), height (centimeter) and surgery duration of the patients in both groups were recorded. Likert evaluation test will be applied for parental satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No